CLINICAL TRIAL: NCT06628375
Title: Exposure to Endocrine Disruptors and Occurrence of Hypospadias: Toxicological, Environmental and Hormonal Imbalance Study
Brief Title: A Multimodal Study of the Relationship Between Exposure to Endocrine Disruptors and Occurrence of Hypospadias - HYPOLLUT
Acronym: HYPOLLUT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0559
Record Dates: First submitted 2024-09-25; First posted 2024-10-08 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Hypospadias
Keywords: Endocrine-disrupting chemicals; Birth defect; Environment; Hormones minipuberty; Exposome; Toxicology hair
MeSH Terms: conditions — Hypospadias; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A blood sample into 5 ml EDTA tube may also be taken from the child with hypospadias, for a DNA collection.
  The remaining hair sample will be kept to measure new pollutant molecules, depending on scientific advancements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case Group: Biological mother and son with hypospadias
  Interventions: Other: Consultation visit (Visit 1)
- Control Group: Biological mother and son without hypospadias
  Interventions: Other: Consultation visit (Visit 1)

INTERVENTIONS:
Other: Consultation visit (Visit 1) — During visit 1, a pediatric urologist or pediatric endocrinologist will perform a clinical examination to confirm the diagnosis of hypospadias, as a part of routine care. The clinical study investigator will ask to fill out a validated European questionnaire for the exposome and use an occupation/exposure matrix to identify specific atmospheric exposure.
  A hair sample from the biological mother will be taken for toxicological evaluation of substances accumulated during pregnancy.
  From the child, a blood sample will be taken for hormonal evaluation of minipuberty and then, another sample in a 5 ml EDTA tube will be taken for DNA collection.
  Groups: Case Group
Other: Consultation visit (Visit 1) — During visit 1, a pediatric urologist or pediatric endocrinologist will perform a clinical examination to confirm the absence of hypospadias. The clinical study investigator will ask to fill out a validated European questionnaire for the exposome and use an occupation/exposure matrix to identify specific atmospheric exposure.
  A hair sample from the biological mother will be taken for toxicological evaluation of substances accumulated during pregnancy.
  From the child, a blood sample will be taken for hormonal evaluation of minipuberty.
  Groups: Control Group

SUMMARY:
This study aims to demonstrate the impact of Endocrine-Disrupting Chemicals (EDCs) on the risk of hypospadias incidence. It is a multicenter comparative case-control study, involving two groups. The first group consists of biological mothers who have given birth to children with hypospadias (Case Group), while the second group consists of biological mothers who have given birth to children without any malformations (Control Group). Through an integrative approach that combines a direct toxicological study of numerous pollutants present during pregnancy, and a comprehensive exposome assessment using validated tools, this study can significantly enhance our understanding and prevention of this malformation.

DETAILED DESCRIPTION:
Background. Hypospadias is a birth defect of the external genital organs in boys and it ranks the second most common genital malformation in male newborns, following cryptorchidism. Its prevalence is increasing in certain global regions, with an estimated rate of 3.8 cases per 1000 male births. To date, the exact cause of hypospadias remains unknown, however genetic, hormonal, and environmental factors are likely involved. Medical and surgical treatment may be necessary. Furthermore, hypospadias is correlated with fertility issues and is also linked to testicular cancer.

Aim. After ruling out hypospadias with a genetic cause, the aim of this study is to evaluate any significant differences to environmental endocrine disrupting-chemicals (EDCs) exposure between biological mothers of children with hypospadias and those with children without malformation. It aims to demonstrate that this exposure (professional, occupational, environmental) leads to hormonal changes during the neonatal mini-puberty period.

Methods. This research will be conducted as a multicenter case-control study: mother and son with isolated anterior or middle hypospadias (Case Group) and mother and son without hypospadias (Control Group). The clinical investigator plans to enroll 200 patients.

A single visit will be performed. This consultation is part of the usual follow-up for children in the Case Group, while it is specific to the project for children in the Control Group.

During this visit, the investigator:

* will establish the diagnosis of hypospadias (for cases) or absence of genital anomaly (for controls)
* will lead an interview using a questionnaire and a job-exposure matrix to assess EDCs during pregnancy
* will take a hair sample from the mother to measure the substances accumulated during pregnancy
* and finally, will take a blood sample from the child for hormonal evaluation of mini-puberty, and another blood sample from child in the Case Group for analysis and the participation in a DNA collection

ELIGIBILITY:
Non-specific Inclusion Criteria :

* Parents of legal age having signed a free and informed consent for the participation of their child
* Biological mother of a boy aged between 1 and 6 months
* Biological mother with a minimum hair length of 18 cm
* Biological mother who has signed a free and informed consent for her participation
* Biological mother and child affiliated with or beneficiaries of a national health insurance plan
* Biological mother who is fluent in written and spoken French

Specific Inclusion Criteria for Case Group:

- The child has an isolated anterior or middle hypospadias, without any other complex variations of genital development (borderline penile size, unilateral or bilateral cryptorchidism, retractile testes), without malformation syndrome and without identified genetic etiology

Specific Inclusion Criteria for Control Group:

- The child must not present any complex variations in genital development (hypospadias, borderline penis size, unilateral or bilateral cryptorchidism, retractile testes)

Exclusion Criteria:

* Child with another congenital anomaly or malformative syndrome
* Child with an endocrine pathology
* Biological mother or child under legal protection, guardianship, or curatorship
* Biological mother or child in the exclusion period of a previous study
* Biological mother or child included in another clinical study involving a drug

Specific Exclusion Criteria for Case Group:

Biological mother/child pairs if a genetic variant explaining hypospadias is found during genetic analysis.

Min Age: 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Case Group: Biological mother and child with hypospadias Control group: Biological mother and child without hypospadias
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-10-03 (Estimated)

PRIMARY OUTCOMES:
Evaluation of toxic exposure via hair sample analysis | Day 1 (Visit 1)
  An assessment of toxic substance concentrations in maternal hair will evaluate exposure to a wide range of pollutants. The collected hair samples will provide data representing the period from three months before conception to the date of study enrollment.
  The study will analyze 150 chemical substances and measure their concentrations to assess mothers' exposure to these pollutants during pregnancy.

SECONDARY OUTCOMES:
Exposome through validated European questionnaires (QLK4-1999-01422) | Day 1 (Visit 1)
  Evaluation of parents' environmental exposure (exposome) will be conducted using a simplified version of a validated European questionnaire. This approach aims to elucidate potential differences in exposure between case and control groups.
Exposome professionnel | Day 1 (Visit 1)
  Assessment by the job-exposure matrix EDC (Environment disrupting chemicals)
Pollutant dispersion model | Day 1 (Visit 1)
  Examination of atmospheric pollutant concentration measurements and their potential impact on maternal exposure during gestation. This study conducts a comparative analysis between two groups: mothers of affected children (case group) and mothers of unaffected children (control group).
Hormonal analysis by immunoassay principle | Day 1 (Visit 1)
  Measurement of plasma hormone levels of mini-puberty to investigate a correlation between toxicological dosage and endocrine disruption. FSH, LH, AMH and free Testosterone will be measured by Electrochemiluminescence and Inhibin B by ELISA assay. This assessment of a mini-puberty alteration will be carried out by comparing age-based norms and the values of the control group

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas KALFA, Prof, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CRMR DEVGEN CHU Lapeyronnie, Montpellier, Hérault, France

REFERENCES:
- [Background] Ea V, Bergougnoux A, Philibert P, Servant-Fauconnet N, Faure A, Breaud J, Gaspari L, Sultan C, Paris F, Kalfa N. How Far Should We Explore Hypospadias? Next-generation Sequencing Applied to a Large Cohort of Hypospadiac Patients. Eur Urol. 2021 Apr;79(4):507-515. doi: 10.1016/j.eururo.2020.12.036. Epub 2021 Jan 16. PMID 33468338
- [Background] Skakkebaek NE, Rajpert-De Meyts E, Main KM. Testicular dysgenesis syndrome: an increasingly common developmental disorder with environmental aspects. Hum Reprod. 2001 May;16(5):972-8. doi: 10.1093/humrep/16.5.972. PMID 11331648
- [Background] Skarin Nordenvall A, Chen Q, Norrby C, Lundholm C, Frisen L, Nordenstrom A, Almqvist C, Nordenskjold A. Fertility in adult men born with hypospadias: A nationwide register-based cohort study on birthrates, the use of assisted reproductive technologies and infertility. Andrology. 2020 Mar;8(2):372-380. doi: 10.1111/andr.12723. Epub 2019 Nov 20. PMID 31670475
- [Background] Springer A, van den Heijkant M, Baumann S. Worldwide prevalence of hypospadias. J Pediatr Urol. 2016 Jun;12(3):152.e1-7. doi: 10.1016/j.jpurol.2015.12.002. Epub 2015 Dec 31. PMID 26810252
- [Background] Schneuer FJ, Milne E, Jamieson SE, Pereira G, Hansen M, Barker A, Holland AJA, Bower C, Nassar N. Association between male genital anomalies and adult male reproductive disorders: a population-based data linkage study spanning more than 40 years. Lancet Child Adolesc Health. 2018 Oct;2(10):736-743. doi: 10.1016/S2352-4642(18)30254-2. Epub 2018 Aug 30. PMID 30236382
- [Background] Asklund C, Jensen TK, Main KM, Sobotka T, Skakkebaek NE, Jorgensen N. Semen quality, reproductive hormones and fertility of men operated for hypospadias. Int J Androl. 2010 Feb;33(1):80-7. doi: 10.1111/j.1365-2605.2009.00957.x. Epub 2009 Mar 5. PMID 19281491
- [Background] Davis CE Jr, Wiley WB, Faulconer RJ. Necrosis of the female breast complicating oral anticoagulant treatment. Ann Surg. 1972 May;175(5):647-56. doi: 10.1097/00000658-197205000-00004. No abstract available. PMID 5028481
- [Background] Serrano T, Chevrier C, Multigner L, Cordier S, Jegou B. International geographic correlation study of the prevalence of disorders of male reproductive health. Hum Reprod. 2013 Jul;28(7):1974-86. doi: 10.1093/humrep/det111. Epub 2013 May 12. PMID 23670171
- [Background] Cortes D, Thorup JM, Visfeldt J. Cryptorchidism: aspects of fertility and neoplasms. A study including data of 1,335 consecutive boys who underwent testicular biopsy simultaneously with surgery for cryptorchidism. Horm Res. 2001;55(1):21-7. doi: 10.1159/000049959. PMID 11423738
- [Background] Pettersson A, Richiardi L, Nordenskjold A, Kaijser M, Akre O. Age at surgery for undescended testis and risk of testicular cancer. N Engl J Med. 2007 May 3;356(18):1835-41. doi: 10.1056/NEJMoa067588. PMID 17476009
- [Background] Xing JS, Bai ZM. Is testicular dysgenesis syndrome a genetic, endocrine, or environmental disease, or an unexplained reproductive disorder? Life Sci. 2018 Feb 1;194:120-129. doi: 10.1016/j.lfs.2017.11.039. Epub 2017 Nov 26. PMID 29183799
- [Background] Olesen IA, Sonne SB, Hoei-Hansen CE, Rajpert-De Meyts E, Skakkebaek NE. Environment, testicular dysgenesis and carcinoma in situ testis. Best Pract Res Clin Endocrinol Metab. 2007 Sep;21(3):462-78. doi: 10.1016/j.beem.2007.04.002. PMID 17875492
- [Background] Stillman RJ. In utero exposure to diethylstilbestrol: adverse effects on the reproductive tract and reproductive performance and male and female offspring. Am J Obstet Gynecol. 1982 Apr 1;142(7):905-21. doi: 10.1016/s0002-9378(16)32540-6. PMID 6121486
- [Background] Lymperi S, Giwercman A. Endocrine disruptors and testicular function. Metabolism. 2018 Sep;86:79-90. doi: 10.1016/j.metabol.2018.03.022. Epub 2018 Mar 29. PMID 29605435
- [Background] Kalfa N, Paris F, Soyer-Gobillard MO, Daures JP, Sultan C. Prevalence of hypospadias in grandsons of women exposed to diethylstilbestrol during pregnancy: a multigenerational national cohort study. Fertil Steril. 2011 Jun 30;95(8):2574-7. doi: 10.1016/j.fertnstert.2011.02.047. Epub 2011 Apr 2. PMID 21458804
- [Background] Vidaeff AC, Sever LE. In utero exposure to environmental estrogens and male reproductive health: a systematic review of biological and epidemiologic evidence. Reprod Toxicol. 2005 May-Jun;20(1):5-20. doi: 10.1016/j.reprotox.2004.12.015. PMID 15808781
- [Background] Giwercman A, Rylander L, Lundberg Giwercman Y. Influence of endocrine disruptors on human male fertility. Reprod Biomed Online. 2007 Dec;15(6):633-42. doi: 10.1016/s1472-6483(10)60530-5. PMID 18062860
- [Background] Sharpe RM, Skakkebaek NE. Testicular dysgenesis syndrome: mechanistic insights and potential new downstream effects. Fertil Steril. 2008 Feb;89(2 Suppl):e33-8. doi: 10.1016/j.fertnstert.2007.12.026. PMID 18308057
- [Background] Parks LG, Ostby JS, Lambright CR, Abbott BD, Klinefelter GR, Barlow NJ, Gray LE Jr. The plasticizer diethylhexyl phthalate induces malformations by decreasing fetal testosterone synthesis during sexual differentiation in the male rat. Toxicol Sci. 2000 Dec;58(2):339-49. doi: 10.1093/toxsci/58.2.339. PMID 11099646
- [Background] Sharpe RM. The 'oestrogen hypothesis'- where do we stand now? Int J Androl. 2003 Feb;26(1):2-15. doi: 10.1046/j.1365-2605.2003.00367.x. PMID 12534932
- [Background] Nilsson EE, Sadler-Riggleman I, Skinner MK. Environmentally induced epigenetic transgenerational inheritance of disease. Environ Epigenet. 2018 Jul 17;4(2):dvy016. doi: 10.1093/eep/dvy016. eCollection 2018 Apr. PMID 30038800
- [Background] Kalfa N, Paris F, Philibert P, Orsini M, Broussous S, Fauconnet-Servant N, Audran F, Gaspari L, Lehors H, Haddad M, Guys JM, Reynaud R, Alessandrini P, Merrot T, Wagner K, Kurzenne JY, Bastiani F, Breaud J, Valla JS, Lacombe GM, Dobremez E, Zahhaf A, Daures JP, Sultan C. Is Hypospadias Associated with Prenatal Exposure to Endocrine Disruptors? A French Collaborative Controlled Study of a Cohort of 300 Consecutive Children Without Genetic Defect. Eur Urol. 2015 Dec;68(6):1023-30. doi: 10.1016/j.eururo.2015.05.008. Epub 2015 May 23. PMID 26007639
- [Background] Brouwers MM, van Tongeren M, Hirst AA, Bretveld RW, Roeleveld N. Occupational exposure to potential endocrine disruptors: further development of a job exposure matrix. Occup Environ Med. 2009 Sep;66(9):607-14. doi: 10.1136/oem.2008.042184. Epub 2009 Mar 13. PMID 19286684
- [Background] Beranger R, Hardy EM, Dexet C, Guldner L, Zaros C, Nougadere A, Metten MA, Chevrier C, Appenzeller BMR. Multiple pesticide analysis in hair samples of pregnant French women: Results from the ELFE national birth cohort. Environ Int. 2018 Nov;120:43-53. doi: 10.1016/j.envint.2018.07.023. Epub 2018 Jul 29. PMID 30064054
- [Background] Peng FJ, Hardy EM, Beranger R, Mezzache S, Bourokba N, Bastien P, Li J, Zaros C, Chevrier C, Palazzi P, Soeur J, Appenzeller BMR. Human exposure to PCBs, PBDEs and bisphenols revealed by hair analysis: A comparison between two adult female populations in China and France. Environ Pollut. 2020 Dec;267:115425. doi: 10.1016/j.envpol.2020.115425. Epub 2020 Aug 15. PMID 32882460